CLINICAL TRIAL: NCT01858181
Title: A Phase I Study of Subcutaneous Ocaratuzumab (Fab- and Fc-engineered Anti-CD20 Monoclonal Antibody) in Patients With Previously Treated CD20+ B-Cell Malignancies
Brief Title: Phase I Study of Subcutaneous Ocaratuzumab in Patients With Previously Treated CD20+ B-Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mentrik Biotech, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEN-001
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Previously Treated CD20+ B-cell Malignancies
MeSH Terms: interventions — ocaratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): SC ocaratuzumab 40 mg weekly x 4 doses
  Interventions: Biological: ocaratuzumab
- Cohort 2 (Experimental): SC ocaratuzumab 80 mg weekly x 4 doses
  Interventions: Biological: ocaratuzumab
- Cohort 3 (Experimental): SC ocaratuzumab 80 mg weekly x 8 doses
  Interventions: Biological: ocaratuzumab

INTERVENTIONS:
Biological: ocaratuzumab
  Other Names: AME-133v, LY2469298

SUMMARY:
Ocaratuzumab is a third-generation, fully humanized IgG1 monoclonal antibody (mAb) targeting the CD20 surface marker on normal and malignant B lymphocytes. It has been optimized for an increased binding for CD20 and an enhanced antibody dependent cell medicated cytotoxicity (ADCC) effector function.

A previous phase I/II study of intravenously (IV) administered ocaratuzumab in refractory/relapsed follicular lymphoma patients has concluded that ocaratuzumab is safe and well-tolerated at doses up to 375mg/ m2 weekly for four weeks.

In this proposed phase I study, ocaratuzumab will be administered subcutaneously to patients with previously treated CD20+ B-cell malignancies. Three dose levels (40 mg weekly x 4 doses, 80 mg weekly x 4 doses, and 80 mg weekly x 8 doses) will be investigated for safety, tolerability, pharmacokinetic, and pharmacodynamic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Histologically confirmed diagnosis of a CD20+ B-cell malignancy;
* Received at least one prior treatment regimen;historically documented CD20-positivity is acceptable;
* Appropriate for single agent study drug therapy as prescribed by this protocol;
* ECOG performance status 0 to 2;
* Adequate hematopoietic, renal, and hepatic functions defined as:

  * Absolute neutrophil count greater than 1000 /mm³
  * Platelet count greater than 75,000/mm³
  * Hemoglobin greater than 8.5 g/dL
  * Serum creatinine ≤ 1.5x upper limit of normal
  * AST, ALT, and total bilirubin ≤ 3x upper limit of normal;
* Ability to understand and the willingness to sign a written informed consent document;
* Life expectancy of 6 months or greater.

Exclusion Criteria:

* Anti-CD20 therapy within 4 weeks of enrollment;
* Systemic chemotherapy or immunotherapy within 14 days of enrollment;
* Chronic systemic steroid therapy defined as prednisone or equivalent 10 mg/day or greater;
* Systemic cytotoxic or immunosuppressive therapy to be administered concomitantly while participating on this study;
* Active infection, chronic or severe infection requiring ongoing antimicrobial therapy.
* Positivity for hepatitis B (defined as HepBs Antigen +), hepatitis C (defined as HepC Antibody +), or HIV; HIV positive patients on antiretroviral therapy will be excluded;
* History of allergic reactions attributed to compounds of similar chemical or biologic composition;
* Significant cardiac disease (New York Heart Association classes III or IV) or unstable angina despite medication;
* Women who are pregnant or breast-feeding;
* Women of child bearing potential who are unwilling to use effective contraception for the duration of the study drug administration and 6 months after final dose of drug is administered;
* Psychiatric illness/social situations that would limit compliance with study requirements;
* Participation in other investigational studies while enrolled on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters following SC ocaratuzumab administration such as area under the curve, maximum serum drug concentration, and elimination half life | Every office visit throughout the study for up to 12 months
Pharmacodynamic profile of B-cell depletion and re-population as measured by CD19+ peripheral blood B lymphocyte count | Baseline, day 1 and 8, 1 mon, 3 mon, 6 mon, and 12 mon post-treatment

SECONDARY OUTCOMES:
Safety and tolerability of SC ocaratuzumab administration as described by the incidence of adverse events such as local injection site reactions or laboratory abnormalities | Every office visit throughout the study for up to 12 months
Immunogenicity as measured by the incidence, titre of human anti-human antibody (HAHA) immune response | Baseline, 1 mon, 2 mon, 3 mon, 6 mon, and 12 mon post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universtity of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Forero-Torres A, de Vos S, Pohlman BL, Pashkevich M, Cronier DM, Dang NH, Carpenter SP, Allan BW, Nelson JG, Slapak CA, Smith MR, Link BK, Wooldridge JE, Ganjoo KN. Results of a phase 1 study of AME-133v (LY2469298), an Fc-engineered humanized monoclonal anti-CD20 antibody, in FcgammaRIIIa-genotyped patients with previously treated follicular lymphoma. Clin Cancer Res. 2012 Mar 1;18(5):1395-403. doi: 10.1158/1078-0432.CCR-11-0850. Epub 2012 Jan 5. PMID 22223529
- [Background] Tobinai K, Ogura M, Kobayashi Y, Uchida T, Watanabe T, Oyama T, Maruyama D, Suzuki T, Mori M, Kasai M, Cronier D, Wooldridge JE, Koshiji M. Phase I study of LY2469298, an Fc-engineered humanized anti-CD20 antibody, in patients with relapsed or refractory follicular lymphoma. Cancer Sci. 2011 Feb;102(2):432-8. doi: 10.1111/j.1349-7006.2010.01809.x. Epub 2011 Jan 12. PMID 21205069